CLINICAL TRIAL: NCT01654471
Title: Validation of the Korean Version of the Walking Impairment Questionnaire in Patients With Peripheral Arterial Disease
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Principal Investigator, Seung-Kee Min, Professor, Seoul National University Hospital
Other Study IDs: WIQ-SNU
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: Walking Impairment Questionnaire; Peripheral arterial occlusive disease; Korean version
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Medical treatment: only medical treatment (regardless of the kinds of medicine)
- Surgical or endovascular treatemnt group: patients underwent surgery or endovascular therapy

SUMMARY:
The aim of the study is to validate the Korean version of Walking Impairment Questionnaire in patients with peripheral arterial occlusive disease.

DETAILED DESCRIPTION:
First, the original version of WIQ will be translated into Korean, then it will be translated into English, again. The translated version will be sent to the original author to compare with the original version. After correcting, the Korean version will be completed.

The patients with peripheral arterial disease will fill in the Korean version of WIQ before starting treatments. Baseline results of arterial function test, toe-brachial index and treadmill test will be recorded. Three months later, the patients will complete the questionnaire again. Arterial function test, toe-brachial index and treadmill test also will be taken again after treatment and the correlation of WIQ and other exams will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 19~ 80 years
* claudication
* Ankle brachial index < 0.9 or TBI < 0.7 (in patients with DM and ABI higher than 1.3)
* patients who can complete the treadmill test (slope 12%, 2.4km/hr)

Exclusion Criteria:

* critical limb ischemia
* Ankle pressure < 40mmHg
* claudication due to other causes (i.e. spinal stenosis, arthritis, etc)
* patients with high risk of coronary artery syndrome during treadmill test

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral arterial disease
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2012-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Reproducibility of Korean version Walking Impairment Questionnaire | One month
  To test reliatbility of WIQ Korean ver., reproducibility of the test was assessed by test-retest procedure of the baseline and 1month afterwards (intraclass correlation coefficient)
Correlation of WIQ score improvement and change in ABI and treadmill test results | 3 months
  Correlation between changes in WIQ score and changes in ABI or treadmill test results (before and after surgical / radiological or pharmacological intervention) were assessed by Pearson's correlation test

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea